CLINICAL TRIAL: NCT01194609
Title: A Pilot Study of Radiation-Immune Cell Combination Therapy in Recurrent or Persistent Cervical Cancer
Brief Title: A Pilot Study of Radiation-Immune Cell Combination Therapy in Cervical Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No further enrollment after two patients
Sponsor: Korea Cancer Center Hospital (Other)
Responsible Party: Principal Investigator, Sang-Young Ryu, A staff at department of obstetrics and gynecology, Korea Cancer Center Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RadImmune Cx-1001
Record Dates: First submitted 2010-09-02; First posted 2010-09-03 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-05

CONDITIONS: Uterine Cervical Neoplasms
Keywords: Low dose radiation; Adoptive immune cell therapy; Cervical cancer; Pilot study
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Radiation; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Low dose radiation, Immune cell therapy (Experimental): Combination treatment of low-dose radiation 20cGy every 3 weeks three times and autologous immune cell therapy 2 consecutive weeks 3 times every 3 weeks
  Interventions: Biological: Immune cell; Radiation: Low dose radiation

INTERVENTIONS:
Biological: Immune cell — InnoLak two consecutive weeks every 3 weeks for 3 times
  Other Names: InnoLAK
Radiation: Low dose radiation — 20cGy whole body radiation every three weeks for three times
  Other Names: Whole body radiation

SUMMARY:
Among the immune cell therapy, autologous adoptive immune cell therapy is a method to transfer the immune cells derived from peripheral white blood cells and expanded and stimulated with various cytokines and tumor specific antigens in cancer patients. Recently, the low-dose radiation is known to increase the immune response in many human cancer patients. In a clinical trial, 70% response rate with combination of low-dose radiation and adoptive immune cell therapy was reported in recurrent melanoma patients. This study is to investigate the feasibility of combination of low-dose radiation and autologous immune cell therapy in recurrent cervical cancer which is resistant to conventional palliative treatment.

DETAILED DESCRIPTION:
Immune cell therapy is considered one of the most promising anti-cancer strategy in many human cancers. Compared to the destructive methods such as surgery, radiation, and chemotherapy, anti-cancer immune therapy is safer and less toxic method in the treatment of human cancer patients.

Among the immune cell therapy, autologous adoptive immune cell therapy is a method to transfer the immune cells derived from peripheral white blood cells and expanded and stimulated with various cytokines and tumor specific antigens in cancer patients. Recent development of the technique to expand immune cells ex vivo make autologous adoptive immune cell therapy much more feasible and popular. However, immune cell therapy showed response of below 10% currently in several clinical trials. The reason of poor response is that the adopted immune cells have to overcome the highly immune compromised environment in advanced or recurrent cancer patients.

The low-dose radiation, defined as the radiation below the therapeutic dose range, is known to increase the immune response in many human cancer patients. Despite the exact mechanism is not well known, the 'danger signal' and the decrease of T-regulatory cells by low-dose radiation are the possible mechanism of enhanced immunity by low-dose radiation. So, the combination of low-dose radiation and immune cell therapy can be a attractive strategy to recurrent or advanced cancer patients who are resistant to conventional treatment.

A challenging clinical trial performed in recurrent melanoma cancers, Dr. Rosenverg reported around 70% response rate with combination of low-dose radiation and adoptive immune cell therapy. However, the feasibility of combination of low-dose radiation and immune cell therapy is still unknown in many human cancers.

This study is to investigate the feasibility of combination of low-dose radiation and autologous immune cell therapy in recurrent cervical cancer which is resistant to conventional palliative treatment. The cervical cancer, highly responsive to radiation, becomes resistant to radiation in case of recurrent disease. We hypothetize that if the low-dose radiation can reverse the immune compromised environment, adoptive immune cells derived from the autologous peripheral blood immune cells will be highly effective in recurrent cervical cancers.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have signed an approved informed consent and authorization permitting release of personal health information.
2. Age 18-75 years
3. Pathologically proven recurrent or persistent cervical cancer patients resistant to conventional palliative chemotherapy or radiation therapy

   1. Persistent tumor more than 1cm after initial chemoradiation or radiation therapy
   2. Persistent tumor more than 1cm after chemoradiation, radiation or chemotherapy in recurrent cervical cancer
   3. Metastatic cervical cancer to lung resistant to conventional chemotherapy
4. ECOG performance status 0, 1, 2.
5. Expected survival more than 3 months
6. Patients must have adequate:

   Hematologic function: ANC ≥ 1,500/mcl, Hemoglobin >10g/dL, platelets ≥ 100,000/mcl Renal function: creatinine ≤ 1.5 x ULN Hepatic function: AST, ALT ≤ 1.5 x ULN,
7. More than 3 weeks from the last day of previous chemotherapy or radiation

Exclusion Criteria:

1. Patients with immune disease or auto-immune disease (ex. rheumatoid arthritis, SLE, immune vasculitis, IDDM)
2. Immune deficiency disease
3. Cancers other than cervical cancer within 5 years
4. Acute myocardial infarction, uncontrolled hypertension
5. Severe allergic disease
6. Severe psychotic disease
7. Those who can be a candidate for curative surgery

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-09; Primary Completion 2011-09 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Response rate | 12months
  Response rate according to RECIST criteria for 12 months

SECONDARY OUTCOMES:
Toxicity | 12months
  Toxcity according to CTCSEver4.0

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Young Ryu, MD, Principal Investigator — Korea Institute of Radiological & Medical Sciences
Locations (1):
- Sang-Young Ryu, Seoul, Nowon-Gu, South Korea